CLINICAL TRIAL: NCT07200804
Title: Exploring the Relationship Between Serum Vitamin D and Atherosclerosis in Hemodialysis Patients: A Cross-sectional Study
Brief Title: Relationship Between Serum Vitamin D and Atherosclerosis in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Hassan, Assistant Professor of Internal Medicine and Nephrology, Faculty of Medicine, Ain shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: FMASU MSO 2/2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Serum; Vitamin D; Atherosclerosis; Hemodialysis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients with normal carotid intima-media thickness (CIMT).
  Interventions: Diagnostic Test: Measurement of Serum Vitamin D Level
- Group B: Patients with increased carotid intima-media thickness (CIMT).
  Interventions: Other: Measurement of Carotid Intima-Media Thickness

INTERVENTIONS:
Diagnostic Test: Measurement of Serum Vitamin D Level — Vitamin D is made of two types, named ergocalciferol (vitamin D2) and cholecalciferol (vitamin D3). Vitamin D2 is produced by converting ergosterol, a fungi and plants sterol, when it is exposed to light from the sun. Vitamin D3 is made differently, as it is formed in animal skin such as human skin with the help of 7-dehydrocholesterol when the skin is exposed to sunlight (UVB radiation).
  Groups: Group A
Other: Measurement of Carotid Intima-Media Thickness — Samples were collected by measuring the carotid intima-media thickness (CIMT) with a Mind ray Real time ultrasound scanner DC-6 doppler machine that has a probe at a frequency of 7.5 MHz. The measurement was done from three different sites each 1 cm proximal to the carotid bulb. The average of three values was taken to determine the final value. If CIMT > 0.8 mm, it was defined as thickened. The measurements adhered to the Mannheim CIMT Consensus (2004-2006)
  Groups: Group B

SUMMARY:
The study aimed to check if there is a link between good vitamin D levels in the blood and subclinical atherosclerosis in people on hemodialysis.

DETAILED DESCRIPTION:
Hemodialysis patients with End-Stage Renal Disease (ESRD) face a significantly elevated risk of cardiovascular disease (CVD) due to a complex interplay of factors. A 30-year-old HD patient faces a cardiovascular mortality risk equivalent to that of an 80-year-old in the general population, emphasizing the accelerated aging of the cardiovascular system in ESRD.

Vitamin D may reduce inflammation and modulate immunity, lowering hypertension and dyslipidemia risks and possibly reversing vascular calcification. However, excessive supplementation can cause hypercalcemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease (ESRD) who had been on maintenance hemodialysis for at least 6 months.
* Age of 18 years or older.
* Patients receiving three weekly dialysis sessions using a bicarbonate-based dialysate with anticoagulants.

Exclusion Criteria:

* Patients with active infections, malignancies, autoimmune diseases, or pre-existing cardiovascular conditions.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present cross-sectional study was carried out on 90 patients with ESRD undergoing hemodialysis at Ain Shams University or the National Institute of Nephrology and Urology from June 2021 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation between Serum Vitamin D and Atherosclerosis | Immediately post-procedure (Up to 1 hour)
  Correlation between Serum Vitamin D and Atherosclerosis was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.